CLINICAL TRIAL: NCT04540705
Title: A Phase 1 Study to Compare Bempegaldesleukin Combined With Nivolumab and Tyrosine Kinase Inhibitor (TKI) to Nivolumab and TKI Alone in Participants With Previously Untreated Advanced or Metastatic Renal Cell Carcinoma (mRCC) (PIVOT IO 011)
Brief Title: A Study to Compare Bempegaldesleukin (BEMPEG: NKTR-214) Combined With Nivolumab and Tyrosine Kinase Inhibitor (TKI) to Nivolumab and TKI Alone in Participants With Previously Untreated Kidney Cancer That is Advanced or Has Spread
Acronym: PIVOT IO 011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA045-011; 2018-003200-39 (EudraCT Number); 18-214-15 (Other: Nektar Therapeutics)
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Renal Cell Carcinoma
Keywords: NKTR-214; nivolumab; bempeg
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Axitinib; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1A (Part 1): Nivolumab + Axitinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Axitinib
- Part 1B (Part 1): Nivolumab + Cabozantinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Cabozantinib

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO
Drug: Axitinib — Specified dose on specified days
  Other Names: INLYTA
  Arms: Part 1A (Part 1): Nivolumab + Axitinib
Drug: Cabozantinib — Specified dose on specified days
  Other Names: Cabometyx
  Arms: Part 1B (Part 1): Nivolumab + Cabozantinib

SUMMARY:
The purpose of this study is in Part 1, to determine the safety of nivolumab, bempegaldesleukin (BEMPEG: NKTR-214), and Tyrosine Kinase Inhibitor (TKI) combination.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of renal cell carcinoma (RCC) with clear cell component including participants who may also have sarcomatoid features
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer (AJCC) Stage 4) RCC
* No prior systemic therapy, including prior PD-L1 therapy, for RCC is allowed with the following exception:

  i) One prior adjuvant or neoadjuvant therapy for completely resectable RCC is allowed. Therapy must have included an agent that targets vascular endothelial growth factor (VEGF) pathway or VEGF receptors and recurrence must have occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy
* Life Expectancy ≥ 12 weeks
* Karnofsky Performance Status (KPS) of at least 70%
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria
* Males and females must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Active CNS brain metastases or leptomeningeal metastases
* Active, known or suspected autoimmune disease
* Inadequately treated adrenal insufficiency
* History of pulmonary embolism (PE), deep vein thrombosis (DVT), or prior clinically significant venous or non-CVA/TIA arterial thromboembolic event (eg, internal jugular vein thrombosis) within 3 months prior to treatment assignment (Part 1) and randomization (Part 2)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) by severity (Part 1) | Up to 2.5 years
Incidence of serious adverse events (SAEs) (Part 1) | Up to 2.5 years
Incidence of dose-limiting toxicities (DLTs) (Part 1) | Up to 2.5 years
Incidence of AEs leading to discontinuation (Part 1) | Up to 5 years
Incidence of immune-mediated adverse events (imAEs) (Part 1) | Up to 5 years
Incidence of changes in clinical laboratory results by severity: Hematology tests (Part 1) | Up to 2.5 years
Incidence of changes in clinical laboratory results by severity: Clinical Chemistry tests (Part 1) | Up to 2.5 years
Incidence of changes in clinical laboratory results by severity: Urinalysis tests (Part 1) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (8):
  - Local Institution - 0005, Springdale, Arkansas
  - Local Institution, Louisville, Kentucky
  - Local Institution - 0001, St Louis, Missouri
  - Local Institution - 0009, New York, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Nashville, Tennessee
  - Local Institution - 0014, Houston, Texas
  - Local Institution - 0007, Seattle, Washington
- Argentina (4):
  - Local Institution - 0025, Mar del Plata, Buenos Aires
  - Local Institution - 0075, Río Cuarto, Córdoba Province
  - Local Institution - 0026, Buenos Aires
  - Local Institution - 0024, San Juan
- Brazil (6):
  - Local Institution - 0030, Belo Horizonte, Minas Gerais
  - Local Institution - 0035, Curitiba, Paraná
  - Local Institution - 0028, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0036, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0032, Barretos, São Paulo
  - Local Institution - 0029, São José do Rio Preto, São Paulo
- Canada (4):
  - Local Institution - 0056, Edmonton, Alberta
  - Local Institution - 0015, Vancouver, British Columbia
  - Local Institution - 0022, St. John's, Newfoundland and Labrador
  - Local Institution - 0008, Toronto, Ontario
- Local Institution - 0079, Marseille, France
- Germany (6):
  - Local Institution - 0042, Essen
  - Local Institution - 0045, Hanover
  - Local Institution - 0040, Jena
  - Local Institution - 0044, Munich
  - Local Institution - 0041, Nuremberg
  - Local Institution - 0046, Würzburg
- Mexico (4):
  - Local Institution - 0050, Zapopan, Jalisco
  - Local Institution - 0048, Mexico City, Mexico City
  - Local Institution - 0049, Monterrey, Nuevo León
  - Local Institution - 0055, Querétaro
- Russia (6):
  - Local Institution - 0059, Moscow
  - Local Institution - 0052, Moscow
  - Local Institution - 0087, Moscow
  - Local Institution - 0051, Novosibirsk
  - Local Institution - 0085, Omsk
  - Local Institution - 0058, Saint Petersburg

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04540705.html